CLINICAL TRIAL: NCT03768063
Title: An Open Label, Multicenter Extension Study in Patients Previously Enrolled in a Genentech and/or F. Hoffmann-La Roche Ltd Sponsored Atezolizumab Study (IMbrella B)
Brief Title: A Study in Patients Previously Enrolled in a Genentech and/or F. Hoffmann-La Roche Ltd Sponsored Atezolizumab Study
Acronym: IMbrella B
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO40729; 2023-506184-34-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2018-11-30; First posted 2018-12-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; Bevacizumab; alectinib; cobimetinib; Vemurafenib; venetoclax; enzalutamide; pembrolizumab; Sunitinib; niraparib; cabozantinib; Pemetrexed; Paclitaxel; emactuzumab; rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atezolizumab Monotherapy (Experimental): Participants will receive atezolizumab by intravenous infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab
- Combined Agents with Atezolizumab (Experimental): Participants will receive treatment of atezolizumab with combined agent(s) as directed per the parent study. Participants will receive agent(s) in combination with atezolizumab at the same dose and schedule, and with the same administration guidelines that were in effect at the time of participant discontinuation from the parent study.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Alectinib; Drug: Cobimetinib; Drug: Vemurafenib; Drug: FAP IL2V; Drug: Venetoclax; Drug: Enzalutamide; Drug: Niraparib; Drug: Cabozantinib; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Emactuzumab; Drug: Rucaparib
- Comparator Treatment (Active Comparator): Participants will receive comparator treatment administration as directed per the parent study. Participants will receive comparator treatment at the same dose and schedule, and with the same administration guidelines that were in effect at the time of participant discontinuation from the parent study.
  Interventions: Drug: Cobimetinib; Drug: Vemurafenib; Drug: Venetoclax; Drug: Enzalutamide; Drug: Pembrolizumab; Drug: Sunitinib; Drug: Niraparib; Drug: Pemetrexed; Drug: Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as a monotherapy or atezolizumab with other agent(s) as per parent protocol. Dosing regimen will continue in accordance with the parent study or at equivalent dose (if applicable) and at the same schedule as the parent study, or switch to a fixed atezolizumab dose of 1200 mg every 3 weeks (Q3W).
  Other Names: Tecentriq
  Arms: Atezolizumab Monotherapy; Combined Agents with Atezolizumab
Drug: Bevacizumab — Bevacizumab will be administered as directed per the parent study.
  Other Names: Avastin
  Arms: Combined Agents with Atezolizumab
Drug: Alectinib — Alectinib will be administered as directed per the parent study.
  Other Names: Alecensa
  Arms: Combined Agents with Atezolizumab
Drug: Cobimetinib — Cobimetinib will be administered as directed per the parent study.
  Other Names: Cotellic
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Vemurafenib — Vemurafenib will be administered as directed per the parent study.
  Other Names: Zelboraf
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: FAP IL2V — FAP IL2V will be administered as directed per the parent study.
  Other Names: simlukafusp alfa
  Arms: Combined Agents with Atezolizumab
Drug: Venetoclax — Venetoclax will be administered as directed per the parent study.
  Other Names: Venclexta
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Enzalutamide — Enzalutamide will be administered as directed per the parent study.
  Other Names: Xtandi
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Pembrolizumab — Pembrolizumab will be administered as directed per the parent study.
  Other Names: Keytruda
  Arms: Comparator Treatment
Drug: Sunitinib — Sunitinib will be administered as directed per the parent study.
  Other Names: Sutent
  Arms: Comparator Treatment
Drug: Niraparib — Niraparib will be administered as directed per the parent study.
  Other Names: Zejula
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Cabozantinib — Cabozantinib will be administered as directed per the parent study.
  Other Names: Cometriq
  Arms: Combined Agents with Atezolizumab
Drug: Pemetrexed — Pemetrexed will be administered as directed per the parent study.
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Paclitaxel — Paclitaxel will be administered as directed per the parent study.
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Emactuzumab — Emactuzumab will be administered as directed per the parent study.
  Arms: Combined Agents with Atezolizumab
Drug: Rucaparib — Rucaparib will be administered as directed per the parent study.
  Arms: Combined Agents with Atezolizumab

SUMMARY:
This is an open-label, multicenter, extension study. Patients who are receiving clinical benefit from atezolizumab monotherapy or atezolizumab in combination with other agent(s) or combination/comparator agent(s) during participation in a Genentech or Roche-sponsored study (the parent study), who are eligible to continue treatment and who do not have access to the study treatment locally, may continue to receive study treatment in this extension study following roll-over from the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for continuing atezolizumab-based therapy at the time of roll-over from the parent study, as per the parent study protocol or
* Eligible for continuing the comparator agent(s) in a Genentech- or Roche-sponsored study as per the parent study protocol, with no access to commercially available comparator agent
* Time between the last dose of treatment received in parent study and first dose in extension study is no longer than the interruption period allowed in the parent study. First dose of study treatment in this extension study will be received within 7 days of the treatment interruption window allowed by the parent study
* Continue to benefit from atezolizumab-based study treatment or from the comparator at the time of roll-over from the parent study as assessed by the investigator
* Negative serum pregnancy test within 7 days prior to start of study treatment in women of childbearing potential
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Meet any of the study treatment discontinuation criteria specified in the parent study at the time of enrollment in this extension study
* Study treatment or comparator agent is commercially marketed in the patient's country for the patient-specific disease and is accessible to the patient
* Treatment with any anti-cancer treatment during the time between last treatment in the parent study and the first dose of study treatment in this extension study
* Permanent discontinuation of atezolizumab for any reason during the parent study or during the time between last treatment in the parent study and the first dose of study treatment in this extension study (if applicable). Exception: Participants who permanently discontinued atezolizumab from parent studies that permit participants to continue treatment with the combination agent(s) alone after permanently discontinuing atezolizumab are eligible to enroll in this study.
* Ongoing serious adverse event(s) that has not resolved to baseline level or Grade ≤1 from the parent study or during the time between the last treatment in the parent study and the first dose of study treatment in this extension study
* Any condition that, in the opinion of the investigator, would interfere with the interpretation of patient safety or place the patient at high risk for treatment-related complications
* Concurrent participation in any therapeutic clinical trial (other than the parent study)
* Pregnant or lactating, or intending to become pregnant during this extension study and for the period after the last dose of study treatment specified in the designated referenced safety information (RSI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2028-07-05 (Estimated); Study Completion 2028-07-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Continued Access to Atezolizumab-Based Therapy and/or Comparator Agent(s) | Day 1 up to maximum 10 years

SECONDARY OUTCOMES:
Percentage of Participants With Serious Adverse Events (SAEs) According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | Day 1 up to 90 days after last dose of study treatment (last dose=until clinical benefit or until death, withdrawal of consent, unacceptable toxicity, pregnancy, non-compliance, or termination by Sponsor, whichever occurs first) (up to maximum 10 years)
Percentage of Participants With Adverse Events of Special Interest Determined According to NCI CTCAE Version 5.0 | Day 1 up to 90 days after last dose of study treatment (last dose=until clinical benefit or until death, withdrawal of consent, unacceptable toxicity, pregnancy, non-compliance, or termination by Sponsor, whichever occurs first) (up to maximum 10 years)
Treatment Duration | Day 1 up to 90 days after last dose of study treatment (last dose=until clinical benefit or until death, withdrawal of consent, unacceptable toxicity, pregnancy, non-compliance, or termination by Sponsor, whichever occurs first) (up to maximum 10 years)
Total Dose Received | Day 1 up to 90 days after last dose of study treatment (last dose=until clinical benefit or until death, withdrawal of consent, unacceptable toxicity, pregnancy, non-compliance, or termination by Sponsor, whichever occurs first) (up to maximum 10 years)
Number of Treatment Cycles | Day 1 up to 90 days after last dose of study treatment (last dose=until clinical benefit or until death, withdrawal of consent, unacceptable toxicity, pregnancy, non-compliance, or termination by Sponsor, whichever occurs first) (up to maximum 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (86):
- United States (8):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University School Of Medicine, Trumbull, Connecticut
  - Advent Health Orlando, Maitland, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Carolina BioOncology Institute, PLCC, Huntersville, North Carolina
  - St. Luke's Cancer Care Associates, Bethlehem, Pennsylvania
  - University of Texas Health Sciences Center in San Antonio, San Antonio, Texas
- St Vincent'S Hospital, Darlinghurst, New South Wales, Australia
- Belgium (3):
  - UZ Leuven, Leuven, Flemish Brabant
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
- Brazil (2):
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
- Multiprofile Hospital for Active Treatment Central Onco Hospital OOD, Plovdiv, Bulgaria
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Masaryk?v onkologický ústav, Brno, Czechia
- Rigshospitalet, København Ø, Denmark
- France (5):
  - CHU Angers, Angers, Pays de la Loire Region
  - Centre Antoine Lacassagne, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - hopital de la Timone, Marseille
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Germany (13):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Krankenhaus Barmherzige Bruder Regensburg, Regensburg, Bavaria
  - Universitätsklinikum Schleswig-Holstein;Campus Lübeck, Lübeck, Schleswig-Holstein
  - Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios-Fachklinik Muenchen-Gauting, Gauting
  - SRH Wald-Klinikum Gera, Gera
  - HOPA MVZ GmbH, Hamburg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Universitaetsklinikum Muenster, Münster
  - Universitaets-Hautklinik Tuebingen, Tübingen
  - Universitaettsklinikum Tübingen, Tübingen
  - Universitätsklinik Tübingen, Tübingen
- Greece (3):
  - Metropolitan Hospital, Piraeus, Attica
  - Laiko General Hospital Athen, Athens
  - Anticancer Hospital Ag. Savas, Athens
- Grupo Angeles, Guatemala City, Guatemala
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (2):
  - Orszagos Onkologiai Intezet, Budapest
  - Szegedi Tudományegyetem, Szeged
- Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- Japan (11):
  - Nagoya University Hospital, Aichi
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - University of Tsukuba Hospital, Ibaraki
  - Kanazawa University Hospital, Ishikawa
  - Sendai Kousei Hospital, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka Habikino Medical Center, Osaka
  - NHO Kinki-Chuo Chest Medical Center, Sakaishi
- Phylasis Clinicas Research S de RL de CV, Toluca, Mexico
- Poland (8):
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Pozna?, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Specjalistyczny Podkarpacki O?rodek Onkologiczny, Brzozów
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
  - Narodowy Instytut Onkologii im. Marii Sk?odowskiej-Curie - Pa?stwowy Instytut Badawczy, Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroc?aw
- Romania (4):
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj Napoca, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Centrul de Oncologie Oncohelp, Timișoara
- Russia (3):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - Russian Oncology Research Center n.a. N.N. Blokhin, Moscow, Moscow Oblast
  - P.A. Herzen Oncological Inst., Moscow, Moscow Oblast
- University Hospital Bratislava, Bratislava, Slovakia
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University College of Medicine, Liver Research Institute, Seoul
- Spain (3):
  - Hospital Universitario Quiron Dexeus, Barcelona
  - Clinica Universidad de Navarra-Madrid, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
- Faculty of Med. Siriraj Hosp., Bangkok, Thailand
- Ukraine (5):
  - Communal Non profit Enterprise Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - National Cancer Institute MOH of Ukraine, Kiev
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs?k Regional Council, Kryvyi Rih
  - Volyn Regional Oncology Dispensary, Lutsk
  - Regional Municipal Institution Sumy Regional Clinical Oncology Dispensary, Sumy

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing